CLINICAL TRIAL: NCT00114556
Title: The Effect Of The Bisphosphonate, Zoledronic Acid, On Bone Density In Liver Transplant Patients - A Prospective, Randomised, Controlled Clinical Trial
Brief Title: The Effect of Zoledronic Acid on Bone Density in Liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CZOL446 AU02
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2004-12

CONDITIONS: Osteoporosis; Liver Transplantation; Fractures
Keywords: osteoporosis; liver transplantation
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
Following liver transplantation, rapid bone loss occurs, particularly within the first 6 months post-transplant. This may be associated with fractures, most notable vertebral. The ability to assess osteoporosis therapies in this system may provide useful information for osteoporosis management in general.

Hypotheses:

1. That treatment with the bisphosphonate, zoledronate, at the time of liver transplantation and at 1 month post-transplantation will prevent the early transplant-related bone loss (measured by bone densitometry and biochemical bone markers at 3 months) seen in patients who are not treated with a bisphosphonate
2. That continuing treatment with zoledronate at 3 monthly intervals for a total duration of 12 months will result in further improvements in bone density beyond that seen at 3 months
3. That calcium and vitamin D (vit D) supplementation of liver transplant patients does not prevent marked bone loss following transplantation.

DETAILED DESCRIPTION:
This study is a prospective, randomised, double-blind, placebo-controlled clinical trial in liver transplant patients comparing therapy with the bisphosphonate, zoledronate, to patients who do not receive bisphosphonate therapy. All groups will receive calcium and vit D supplementation from the time patients are listed for transplantation and for 12 months post-transplantation. Recruited subjects will be 17 years or older (ie adult in terms of consent requirements).

The study groups comprise:

Group 1: Zoledronate plus calcium and vit D supplementation

Zoledronate 4 mg will be administered by intravenous infusion (details below) at baseline (within 72 h of liver transplantation), followed by zoledronate 4 mg infused as outlined below at 1, 3, 6 and 9 months post-transplantation PLUS calcium 600mg daily (Caltrate, one tablet) and ergocalciferol 1000 IU daily (Ostelin, one capsule) for 12 months post-transplantation.

Group 2: Placebo plus calcium and vit D supplementation

Placebo will consist of 50 ml N/Saline infused over 15 minutes as for the zoledronate regime PLUS calcium 600mg daily (Caltrate, one tablet) and ergocalciferol 1000 IU daily (Ostelin, one capsule). Patients with low vitamin D levels (<60 nmol/L) and parathyroid hormone (Pth) levels above normal >6.5 should receive ergocalciferol 5000 U daily.

Zoledronate/Placebo Infusion regime

Zoledronate 4 mg will be infused in 100 ml N/Saline over 15 minutes in patients with a creatinine level <1.5 times the upper limit of the normal range (i.e <165 µmol/L). Patients with renal impairment as indicated by a serum creatinine level >1.5 x ULN will be discussed on an individual basis with the Medical Adviser of Novartis. If zoledronate is to be given, an extended infusion time may be used. Renal toxicity has been reported with rapid infusions (5 min) of 8 mg of zoledronate in patients with pre-existing renal failure. Further pharmacokinetic studies in patients with renal failure are being undertaken by Novartis to clarify this area. Zoledronate infusion should be freshly prepared and administered without delay.

The Hospital Pharmacy will be responsible for providing the infusions (zoledronate reconstituted in N/Saline or N/Saline alone), appropriately masked, for both Groups 1 and 2.

Primary Outcome Measures:

1) Bone Density at 3 months post-transplantation

Maximal loss of bone following transplantation is seen by 3 months. Earlier data on bone loss in liver transplant patients from the RPAH unit demonstrated an average of 24% bone loss by 3 months post-transplantation. Prevention of this effect should provide a precise and early measurement of the effect of zoledronate on transplant-related bone loss. Bone density of the hip, spine, and total body will be measured by dual xray absorptiometry (DEXA) at baseline (not more than 6 months prior to liver transplantation), and 3, 6 and 12 months following liver transplantation.

Secondary Outcome Measures:

1. Bone Density at 6 and 12 months post-transplantation

   The BMD assessments at 6 and 12 months will assess further changes in bone density between the treated and control groups beyond those assessed at 3 months.
2. Biochemical Markers of Bone Metabolism

   Biochemical markers of bone formation (osteocalcin and total and bone specific alkaline phosphatase) and bone resorption (urinary collagen cross-links, N-teleopeptide and deoxypyridinoline, as well as serum cross-links, C-teleopeptide) will be assayed in serum/urine collected at baseline, and 1, 3, 6, 9 and 12 months following liver transplantation.
3. Fracture Events Fracture incidence in the RPAH patients has been previously reported as 17% in the first 6 months post-transplantation. The fracture rate is now probably lower due to improvements in immunosuppressive therapy. It is not anticipated that this study will have sufficient power to detect a significant reduction in fractures however fracture events will be recorded, including reduction in height of vertebral bodies at baseline and 12 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 17 years of age

Exclusion Criteria:

* Concurrent treatment, or within the past 12 months, with drugs known to affect bone metabolism
* Hypocalcemia
* Renal impairment (creatinine >1.5x ULN)

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2000-02; Study Completion 2004-08

PRIMARY OUTCOMES:
bone density

SECONDARY OUTCOMES:
bone turnover markers

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey McCaughan, PhD, MB BS, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia
Locations (1):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] McDonald JA, Dunstan CR, Dilworth P, Sherbon K, Sheil AG, Evans RA, McCaughan GW. Bone loss after liver transplantation. Hepatology. 1991 Oct;14(4 Pt 1):613-9. doi: 10.1016/0270-9139(91)90047-y. PMID 1916662
- [Result] Crawford BA, Kam C, Pavlovic J, Byth K, Handelsman DJ, Angus PW, McCaughan GW. Zoledronic acid prevents bone loss after liver transplantation: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2006 Feb 21;144(4):239-48. doi: 10.7326/0003-4819-144-4-200602210-00005. PMID 16490909